CLINICAL TRIAL: NCT02421497
Title: MRI Technical Development and Applications in Kidney Disease
Status: Not yet recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1410M54981
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Diseases; Kidney Transplantation; Dialysis; Cognition Disorders
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cognition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Normal Healthy Volunteer
- Non-CKD Control
- Chronic Kidney Disease (CKD)
- Dialysis Patients
- Renal Transplant Recipients

SUMMARY:
Magnetic resonance imaging (MRI), as a non-invasive and non-contrast enhanced technique, has the potential to improve patient health care and management. The overall objective of proposed project is to:

1. develop, customize, and optimize anatomic and functional MRI methods,
2. explore the use of MRI methods to study CKD and evaluate post-transplant kidneys, and
3. investigate the potential of MRI in the diagnosis, prognosis, and monitoring of the progression of renal dysfunction.

In addition to direct studies of the kidney, brain MRI studies will also be performed to identify the cerebrovascular and cognitive effects of chronic renal function deficiency and medical treatment (e.g. hemodialysis and immunosuppression). The brain and kidneys have similar vascular bed, and both are susceptible to vascular injury, which provides the pathological basis for the widely recognized association of reduced renal function with prevalent cerebrovascular diseases (CVDs) and cognitive impairment (CI). The MRI methods in the brain will be applied to explore the origins for widely observed CVDs and prevalent cognitive impairment (CI) in kidney disease patients.

DETAILED DESCRIPTION:
Specific Aims

The overall objective is to develop and validate MRI methods for the evaluation and monitoring of renal status and associated cerebrovascular effects of renal dysfunction and treatment. The proposed project include two phases: 1) MRI technical development and validation with reproducibility studies; 2) clinical pilot studies with two patient populations (CKD patients and renal transplant recipients) to explore the potential of MRI in evaluating CKD, post-transplantation renal dysfunction and cerebrovascular pathophysiology associated with or induced by reduced kidney function and renal replacement treatment. The ultimate goal is to use MRI as a non-invasive and non-contrast enhanced tool to facilitate the diagnosis and prognosis of renal dysfunction and associated diseases, and to assess the efficacy of therapeutic interventions, and monitor disease progress across time.

Specific Aim 1: Imaging technical development and protocol optimization for renal and cerebral MRI.

The overall goal is to develop, customize and optimize new MRI methods to overcome challenges due to physiological motions and facilitate clinical research studies of renal and cerebral diseases, which will include but not are limited to the following aspects.

Sub-Aim 1.1: Develop imaging methods to improve MRI quality and efficiency for renal disease studies.

Sub-Aim 1.2: Optimize gas-challenge functional MRI protocols to study cerebral and renal vascular endothelial dysfunction.

Sub-Aim 1.3: Evaluate the reproducibility of cerebral and renal MRI methods.

Specific Aim 2: Perform pilot studies to evaluate the potential of MRI in CKD patients and renal transplant recipients.

Sub-Aim 2.1: Evaluate the correspondence of MRI measures with clinical metrics (i.e. eGFR) and routinely assessed cognitive functions from CKD and ESRD patients.

This will be accomplished by performing both cross-sectional and longitudinal studies, which will allow us to evaluate the diagnostic and prognostic potential of these non-invasive imaging methods. The investigators hypothesize that the measurements from cerebral and/or renal MRI can effectively reflect cerebral and/or renal (anatomic and physiological) changes induced by CKD or dialysis treatment.

Sub-Aim 2.2: Investigate the potential of MRI methods in the evaluation of post-transplant kidneys.

This will be accomplished by imaging transplant recipients in three distinct cohorts; those with good allograft function but coming in for routine protocol biopsy, with stable renal function, and with unstable renal function due to post-transplant complications. These patient populations will receive protocol biopsies (i.e. scheduled repeat biopsies) as standard of care; therefore pathologic results will be available for correlation with MRI measures. The investigators hypothesize that MRI methods can be a non-invasive surrogate marker of renal tissue properties and functional changes induced by renal post-transplant dysfunction (e.g. renal rejection) currently only obtained through biopsy.

ELIGIBILITY:
For Specific Aim 1: MRI Technical Development Studies

Inclusion Criteria:

1. Healthy Volunteer

Exclusion Criteria:

1. Ferromagnetic implants
2. Any foreign metal objects in the body
3. History of shrapnel or shot gun injury
4. Cardiac pacemakers
5. Defibrillator
6. Neuronal stimulator
7. Magnetic aneurysm clip
8. Large tattoos on the abdomen or the brain and neck
9. Hip replacement
10. Too large to fit in the magnet (body mass index >= 40, approx.)
11. Severe claustrophobia
12. Women with pregnancy

For Specific Aim 2: Pilot Studies with Patients

Studies for CKD

Inclusion

1. English- speaking as primary language.
2. Age 45 years and older
3. Able to complete an approximately 90 minute cognitive testing battery.
4. Able to sign the informed consent, or allow a caregiver, relative, surrogate, or witness to sign the informed consent if participant is unable to do so.
5. GFR < 90 ml/min/1.73m2

Exclusion

1. Acute psychiatric illness that would impede cognitive testing
2. Active chemical dependence, such as alcohol, narcotics or other drugs
3. Legally blind or unable to complete cognitive tests due to visual loss or deafness
4. Dialysis dependent or renal transplant recipient at time of screening or baseline
5. Chronic obstructive pulmonary disease
6. Severe CI unable to complete the Modified Mini-Mental State Examination [3MSE]

Studies for Renal Transplantation

Inclusion

1. Able to sign the informed consent, or allow a caregiver, relative, surrogate, or witness to sign the informed consent if participant is unable to do so.
2. Age 45 years and older

Exclusion

1. Not on dialysis due to allograft failure
2. Chronic obstructive pulmonary disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study populations vary across specific aims: normal healthy or control volunteers for Specific Aim 1, CKD patients and renal transplant recipients for Specific Aim 2.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2026-03-30 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Correspondence of MRI measures with clinical metrics (i.e. eGFR) and routinely assessed cognitive functions from CKD and ESRD patients. | up to three years
  MRI measures will be evaluated both globally and regionally (e.g. frontal lobe and the hippocampus of the brain, renal cortex and medulla in each and both kidneys). The correlations among MRI measurements, the degree of CKD disease (as evaluated by eGFR) and the severity of cognitive impairment will be assessed using both cross-sectional and longitudinal analyses. Non-parametric analysis approach will be used instead of parametric if appropriate.
The potential of MRI methods in the evaluation of post-transplant kidneys. | Up to three years
  For each region in kidneys (renal cortex and medulla), each MRI measurement from the cross-sectional studies of transplant recipients with stable renal functional will be correlated to the levels of transplant kidney function (e.g. eGFR). Imaging results from transplant recipients with unstable renal function will be compared between patients with and without diagnosed acute rejection, and before and after the acute rejection treatment for patients with positive response.
  Note: For both outcomes, multi-parametric MRI measurements will be used in the evaluation, including but not limited to MRI relaxation times, blood flow and diffusion.

CONTACTS AND LOCATIONS:
Overall Officials: Xiufeng Li, Ph.D., Principal Investigator — Univesity of Minnesota
Locations (1):
- Center for Magnetic Resonance Research, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided